CLINICAL TRIAL: NCT03912116
Title: Adjunctive Use of Amniotic Umbilical Cord Particulate During Total Knee Arthroplasty
Brief Title: Amniotic Umbilical Cord Particulate During Total Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Personnel Changes
Sponsor: BioTissue Holdings, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLARIX- CS007
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis: Joint Replacement Surgery
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amniotic Umbilical Cord Particulate Injection (Experimental): 100mg Amniotic Umbilical Cord Particulate in 8cc saline
  Interventions: Other: CLARIX FLO; Other: Saline
- Saline Injection (Placebo Comparator): 8cc saline
  Interventions: Other: Saline

INTERVENTIONS:
Other: CLARIX FLO — 100mg CLARIX FLO
  Arms: Amniotic Umbilical Cord Particulate Injection
Other: Saline — Saline

SUMMARY:
Total knee arthroplasty (TKA) is the most common joint replacement surgery and its incidence is expected to increase 673% to 3.48 million procedures annually by 2030. After more than 20 years of follow-up data, TKA is confirmed to be an effective treatment for knee osteoarthritis, however, postoperative pain management continues to be a challenge despite advances in surgical techniques and anesthetic practice to minimize discomfort and enhance recovery. This acute post-surgical pain caused by extensive tissue damage and inflammation in TKA leads to restricted post-operative knee range of motion (ROM) and ability to mobilize.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, greater than 18 years of age
2. Primary diagnosis of unilateral osteoarthritis of the knee
3. Scheduled to undergo primary, unilateral TKA
4. ASA physical status 1, 2, or 3

Exclusion Criteria:

1. Patient has concurrent painful physical condition not strictly related to the knee surgery that may require analgesic treatment (such as NSAIDs or opioid) that may confound postsurgical assessments as determined by the investigator
2. Patient on chronic daily narcotic medication for knee pain based on medical history and Florida Prescription Drug Monitoring Program (E-FORCSE)
3. Allergy or contraindication to any of the study medications
4. Patient reported renal impairment based on medical history
5. Bodyweight less than 50 kg (110 pounds) or a body mass index greater than 40 kg/m2
6. History of previous fracture or open surgery on the knee being considered for TKA
7. History of patellar instability, e.g., Valgus deformity
8. History of inflammatory arthropathy (e.g., Rheumatoid arthritis, Lupus, etc.)
9. Use of cryoneurolysis, or cryoanalgesia, including iovera® device (Myoscience, Fremont, CA) on the operative knee within the last 6 months or planned during study duration
10. Any neurologic disorder or psychiatric disorder (e.g., Parkinson's Multiple Sclerosis, etc.) that might impact postsurgical pain or confound postsurgical assessments
11. Planned use of intra-articular steroid injections during the study.
12. Received any local anesthetic within 7 days of the planned TKA procedure aside from those part of the protocol
13. Planned use of potent inhalational agents or peripheral nerve block (e.g., femoral nerve block)
14. Current or planned use of neuraxial (epidural or intrathecal) opioids
15. Received administration of an investigational drug within 30 days prior to study, and/or has planned administration of another investigational product or procedure during participation in this study
16. History of suspected, or known, misuse, abuse, dependence of opioid analgesics, illicit drugs, prescription medicines, or alcohol within the past 2 years
17. Currently pregnant, nursing, or planning to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2019-12-16 (Actual)

PRIMARY OUTCOMES:
Difference in Pain at 2 weeks: visual analog scale | 2 weeks
  Pain assessed using 100mm visual analog scale (0 to 100 worst possible pain)

SECONDARY OUTCOMES:
Difference in Pain at 5-7 days: visual analog scale | 5-7 days
  Pain assessed using 100mm visual analog scale (0 to 100 worst possible pain)
Difference in Patient Satisfaction: Questionnaire | 2 weeks
  Questionnaire ranging from 1 (Very satisfied), 2 (Satisfied), 3 (Neither satisfied nor dissatisfied, 4 (Dissatisfied), and 5 (Very dissatisfied).
Difference in Quality of Life: SF-36 | 2 weeks
  Assessed by SF-36 (0-100 scale with 100 representing no disability)
Difference in Subjective Outcome | 2 weeks
  Oxford Knee Scale (score 0 most severe symptoms to 48 least symptoms)
Difference in pain medication consumption | 2 weeks
  opioid consumption (morphine equivalents)
Difference in range of motion between baseline and 2 weeks | 2 weeks
  degrees the knee joint can move
Length of Hospital Stay | 5 days
Difference in Number of Readmissions | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Orange Park Medical Center, Orange Park, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided